CLINICAL TRIAL: NCT00313898
Title: The Effect of Treatment for ED on Quality of Life and Satisfaction in a Group of Patients Without Prior Complaints of Sexual Dysfunction
Brief Title: Effect of Sildenafil on Quality of Sexual Life in Mild to Normally Sexually Functioning Males
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: viagracommCTIL
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2006-04

CONDITIONS: Erectile Dysfunction
Keywords: quality of sexual life, Mild erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sildenafil (viagra)

SUMMARY:
In clinical practice it is quite common to have sexually active male patients with mild/normal erectile function that are not satisfied with their sexual function. The aim of this study is to evaluate the effect of sildenafil on the quality of sexual function in this group of patients.

The endpoint of this study is to define another, different group of patients that may respond positively to treatment with sildenafil.

DETAILED DESCRIPTION:
This will be a prospective, placebo-controlled, double blind crossover study. One hundred males between 35-70 years of age in good general health will be included. Recruitment of patients will be done through patient referral to the "male sexual dysfunction clinic" at Rambam Medical Center, as well as by other necessary ways for optimal and rapid recruitment (media advertisement, direct contact with primary clinics etc.).

For each patient, the study will terminate after a maximal period of 4 months from initiation and will include 4 visits:

On inclusion (Visit I), a thorough explanation will be given to each patient on the aims and course of the study, as well as a full explanation on dosage, mode of administration, safety and efficacy of Viagra. After reading and signing an informed consent, each patient will be asked to fill a questionnaire regarding his sexual function (IIEF-ED Domain). If the patient fits inclusion criteria, he will be referred to the urologist to initiate the study. On the second encounter (Visit II), medical history and physical exam will be performed. The subject will then fill out 3 questionnaires: IIEF (full version), QVS (quality of sexual life questionnaire) and the SEARS questionnaire. Administration of medication will be performed in a double-blinded crossover fashion. Each patient will be provided, at random either 6 tablets of placebo or Viagra 50mg. The patient will be advised to use them on demand. After consuming all 6 tablets, a third visit will be scheduled. On the third visit (Visit III) each patient will be provided with new IIEF (full version), QVS (quality of sexual life questionnaire), the SEARS questionnaire and an EDITS questionnaire. A few other questions on satisfaction will be asked and recorded (questions on the quality of the erection, duration of intercourse, number of sexual acts per night, frequency of intercourse/week, satisfaction from intercourse etc). Each subject will receive another 6 tablets (Viagra/ placebo). Finally, at the last visit (Visit IV) subjects will again fill out the same questionnaires as on visit III. At the end of the study, double-blind codes will be opened and multi-variant analysis of the data will be performed using chi square and annova.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active males.
* All males between 35-70 years of age that previously have not taken any PDE5 inhibitors.
* A score of 22/30 and above of the International Index of Erectile Function (IIEF) ED domain (questions 1,2,3,4,5,15) .

Exclusion criteria:

* Patients with psychiatric disorders
* Patients with contraindications to sildenafil (patients on nitrate prescription, very low blood pressure, multiple anti-hypertensive medications, allergy to PDE5i, severe renal or hepatic insufficiency etc)
* Patients with a severe coronary artery disease
* Patients with premature ejaculation as their primary problem without a current partner.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
changes in scoring of quality of sexual life questionnaires before vs after treatment

SECONDARY OUTCOMES:
changes in scoring of erectile function domain

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Israel Urology association
Locations (1):
- Rambam Health Care Campus, Haifa, Israel